CLINICAL TRIAL: NCT01367756
Title: A Single Center, Randomized, Double-blind, Parallel-design Study to Investigate the Safety and Tolerability of RO4995819 in Combination With Citalopram Following Oral Administration in Healthy Volunteers
Brief Title: A Study of RO4995819 in Combination With Citalopram in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP25679
Record Dates: First submitted 2011-05-30; First posted 2011-06-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO4995819; Drug: citalopram
- 2 (Placebo Comparator)
  Interventions: Drug: citalopram; Drug: placebo

INTERVENTIONS:
Drug: RO4995819 — multiple oral doses, Days 10-16
  Arms: 1
Drug: citalopram — multiple oral doses, Days 1-16
Drug: placebo — multiple oral doses, Days 10-16
  Arms: 2

SUMMARY:
This randomized, double-blind, parallel-arm study will assess the safety and tolerability of RO4995819 in combination with citalopram in healthy volunteers. Subjects will receive citalopram orally on Days 1-9 and be randomized to receive either RO4995819 orally or placebo in combination with citalopram on Days 10-16. Safety follow-up will be up to Day 58.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy male or female subjects, 18 to 65 years of age inclusive (healthy status defined as absence of evidence of any active or chronic disease)
* Body mass index (BMI) 18.0 to 30.0 kg/m2 inclusive
* Female subjects who are not either surgically sterile or post-menopausal must commit to using a barrier form of contraception in addition to either an intrauterine device or hormonal contraception until at least 5 months after the last dose of study drug
* Male subjects must use a barrier method of contraception throughout the study and for up to 5 months after the last dose of study drug (applies also to surgically sterilized males)
* Willing not to participate in any other clinical trial with an investigational drug for at least 5 months following the last dose of study drug

Exclusion Criteria:

* Pregnant or lactating females
* Suspicion of regular consumption of drug of abuse or positive test for alcohol on Day -2
* Hepatitis B, hepatitis C or HIV infection
* Smokers of >5 cigarettes or equivalent tobacco intake per day
* Any confirmed allergic reaction against any drug, or multiple allergies (non-active hay fever is acceptable)
* Participation in an investigational drug or device study within 3 months prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to 58 days

SECONDARY OUTCOMES:
Effect of multiple doses of RO4995819 on the pharmacokinetics (Cmax, AUC) of citalopram | 17 days
Effect of genetic variants of drug metabolism on pharmacokinetics (Cmax, AUC) of RO4995819 in combination with citalopram | up to 58 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France